CLINICAL TRIAL: NCT00171314
Title: The Use of Zoledronic Acid to Prevent Cancer-treatment Bone Loss in Post-menopausal Women Receiving Adjuvant Letrozole for Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFEM345D2406
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2012-04-11 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-03

CONDITIONS: Breast Cancer
Keywords: breast cancer; letrozole; zoledronic acid; adjuvant; postmenopausal
MeSH Terms: conditions — Breast Neoplasms | interventions — Zoledronic Acid; Letrozole

ARMS (2):
- Upfront Zoledronic Acid (Experimental): Zoledronic acid 4 mg Intravenous (IV) 15 minute infusion every 6 months for 5 years beginning on Day 1. All participants took Letrozole tablets 2.5 mg/day for 5 years beginning on Day 1
  Interventions: Drug: Zoledronic acid; Drug: Letrozole
- Delayed Zoledronic Acid (Experimental): Zoledronic acid 4 mg Intravenous (IV) 15 minute infusion every 6 months beginning when one of the following occurred: BMD T-score <= -2.0 SD at either the lumbar spine or total hip, any clinical fracture unrelated to trauma or an asymptomatic fracture discovered at the Month 36 visit. All participants took Letrozole tablets 2.5 mg/day for 5 years beginning on Day 1
  Interventions: Drug: Zoledronic acid; Drug: Letrozole

INTERVENTIONS:
Drug: Zoledronic acid — Zoledronic acid 4 mg Intravenous (IV)15 minute infusion every 6 months.
  Other Names: ZOL446; Zometa®
Drug: Letrozole — Letrozole tablets 2.5 mg/day/taken orally for 5 years.
  Other Names: Femara®

SUMMARY:
Post-menopausal breast cancer patients will receive letrozole 2.5 mg daily for the treatment of breast cancer and will be randomized to a treatment group to receive either upfront zoledronic acid 4 mg IV 15-minute infusion every 6 months or delayed start zoledronic acid 4 mg IV 15-minute infusion every 6 months. Delayed start zoledronic acid will be initiated when either the Bone Mineral Density T-score is below -2 Standard Deviations at either the lumbar spine or hip or any clinical fracture unrelated to trauma or an asymptomatic fracture discovered at the month 36 scheduled visit. Letrozole 2.5 mg will be given daily for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-IIIa breast cancer
* Postmenopausal
* Recent surgery for breast cancer

Exclusion Criteria:

* Metastatic disease
* Invasive bilateral disease
* Clinical or radiological evidence of existing fracture in spine or hip

Other protocol-defined inclusion / exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 527 (Actual)
Dates: Start 2004-03; Primary Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (49):
- Argentina (2):
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Rosario - Santa Fe
- Belgium (15):
  - Novartis Investigative Site, Aalst
  - Novartis Investigative Site, Anderlecht
  - Novartis Investigative Site, Bonheiden
  - Novartis Investigative Site, Brasschaat
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Hasselt
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Libramont-Chevigny
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Mons
  - Novartis Investigative Site, Ottignies
  - Novartis Investigative Site, Saint Niklaas
  - Novartis Investigative Site, Wilrijk
  - Novartis Investigative Site, Yvoir
- France (8):
  - Novartis Investigative Site, Limoges
  - Novartis Investigative Site, Mougins
  - Novartis Investigative Site, Périgueux
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Saint-Brieuc
  - Novartis Investigative Site, Saint-Herblain
  - Novartis Investigative Site, Toulon
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Italy (9):
  - Novartis Investigative Site, Genova
  - Novartis Investigative Site, Ivrea
  - Novartis Investigative Site, Lecco
  - Novartis Investigative Site, Monteforte Irpino (Av)
  - Novartis Investigative Site, Pietra Ligure
  - Novartis Investigative Site, Roma
  - Novartis Investigative Site, Sassari
  - Novartis Investigative Site, Torino
  - Novartis Investigative Site, Vicenza
- Netherlands (4):
  - Novartis Investigative Site, Eindhoven
  - Novartis Investigative Site, Hoogeveen
  - Novartis Investigative Site, Nijmegen
  - Novartis Investigative Site, The Hague
- Novartis Investigative Site, Riyadh, Saudi Arabia
- South Africa (3):
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Durban
  - Novartis Investigative Site, Johannesburg
- South Korea (3):
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Jeollanam-do
  - Novartis Investigative Site, Seoul
- Spain (4):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Upfront Zoledronic Acid | Delayed Zoledronic Acid
Started | 263 (2 patients in each arm were randomized but not treated.) | 264
Safety Population | 254 (Treatment Actually Received = 251 from "upfront" Arm and 3 from "delayed" Arm) | 269 (Treatment Actually Received = 10 from "upfront" Arm and 259 from "delayed" Arm)
Completed | 172 | 186
Not Completed | 91 | 78
Not completed — Adverse Event | 44 | 41
Not completed — Lack of Efficacy | 19 | 14
Not completed — Withdrawal by Subject | 9 | 6
Not completed — Abnormal Test Procedure Results | 9 | 3
Not completed — Protocol Violation | 3 | 7
Not completed — Administrative Problems | 4 | 3
Not completed — Lost to Follow-up | 1 | 3
Not completed — Death | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Upfront Zoledronic Acid | Delayed Zoledronic Acid | Total
Number analyzed (Participants) | 263 | 264 | 527
Age Continuous [Mean (Standard Deviation); unit: years] | 58.2 (8.19) | 58.4 (7.73) | 58.29 (7.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 263 | 264 | 527
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Lumbar Spine (L2-L4) BMD After 12 Months of Letrozole Therapy
Description: Bone Mineral Density (BMD)is measured by dual energy x-ray absorptiometry (DXA).Percent Change = [(BMD at Visit - BMD at Baseline) / BMD at Baseline] * 100.
Time Frame: From Baseline - 12 months
Population: For the analysis of safety, the safety population for treatment arms were defined by the actual treatment received, rather than the treatment arm assigned by randomization. Participants with observations at baseline and 12 months were included in this analysis.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Upfront Zoledronic Acid | Delayed Zoledronic Acid
Number analyzed (Participants) | 254 | 269
Percent Change | 2.680 (2.8451) | -3.314 (3.9632)

2. Secondary Outcome: Percent Change in Lumbar Spine (L2-L4) BMD at 2 Years, 3 Years, 4 Years and 5 Years
Description: as for outcome 1
Time Frame: From Baseline to Year 2, Year 3, Year 4, Year 5
Population: Analysis of safety:safety population for treatment arms were defined by the actual treatment received, rather than the treatment arm assigned by randomization. "n" in each category indicates participants with data at baseline and each corresponding timepoint.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Upfront Zoledronic Acid | Delayed Zoledronic Acid
Number analyzed (Participants) | 254 | 269
Percent Change
  Year 2 (n=122,142) | 4.136 (3.8182) | -3.924 (4.7442)
  Year 3 (n=119,133) | 4.777 (4.8959) | -4.297 (5.3583)
  Year 4 (n=104, 122) | 5.462 (5.2922) | -4.746 (5.6588)
  Year 5 (n=86, 102) | 6.013 (5.4366) | -4.572 (6.1617)

3. Secondary Outcome: Percent Change in Lumbar Spine (L1-L4) BMD at Year 1, Year 2, Year 3, Year 4 and Year 5
Description: as for outcome 1
Time Frame: From Baseline to Year 1, Year 2, Year 3, Year 4, Year 5
Population: For the analysis of safety, the safety population for treatment arms were defined by the actual treatment received, rather than the treatment arm assigned by randomization.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Upfront Zoledronic Acid | Delayed Zoledronic Acid
Number analyzed (Participants) | 254 | 269
Percent Change
  Year 1 (n=123, 156) | 2.330 (2.7465) | -3.532 (3.7830)
  Year 2 (n=122, 142) | 3.994 (3.6344) | -3.934 (4.7162)
  Year 3 (n=199, 133) | 4.523 (4.5197) | -4.292 (5.2317)
  Year 4 (n=104, 122) | 5.051 (4.9739) | -4.713 (5.4101)
  Year 5 (n=86, 102) | 5.476 (5.0395) | -4.692 (6.0242)

4. Secondary Outcome: Percent Change in Total Hip BMD at Year 1, Year 2, Year 3, Year 4 and Year 5
Description: as for outcome 1
Time Frame: From baseline to Year 1, Year 2, Year 3, Year 4, Year 5
Population: For the analysis of safety, the safety population for treatment arms were defined by the actual treatment received, rather than the treatment arm assigned by randomization. During different time points, participants with observations at that time point were included in the analysis.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Upfront Zoledronic Acid | Delayed Zoledronic Acid
Number analyzed (Participants) | 254 | 269
Percent Change
  Year 1 (n=173, 187) | 1.637 (2.4371) | -1.644 (2.9994)
  Year 2 (n=169, 168) | 2.119 (2.9435) | -2.628 (3.5659)
  Year 3 (n=163, 162) | 1.991 (3.4207) | -3.011 (4.7684)
  Year 4 (n=145, 152) | 2.439 (3.5236) | -3.074 (5.4515)
  Year 5 (n=119, 121) | 2.788 (3.8386) | -4.012 (5.1321)

5. Secondary Outcome: Percentage of Participants With Radiological (Vertebra) Fractures Which Were Not Present at Baseline But Were Present at Year 3
Description: Radiological Fracture at 36 months which was not present at baseline = (new fracture/number participant analyzed)*100. Evaluation of radiological fractures were based on central lab X-ray data. A subject with multiple fractures at the same time or multiple fractures with the same grade is counted only once for that treatment.
Time Frame: Year 3
Population: For the analysis of safety, the safety population for treatment arms were defined by the actual treatment received, rather than the treatment arm assigned by randomization. Participants with observations at Year 3 were included in this analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Upfront Zoledronic Acid | Delayed Zoledronic Acid
Number analyzed (Participants) | 254 | 269
Percentage of Participants | 2.8 | 3.3

ADVERSE EVENTS:
Arm/Group | Upfront Zoledronic Acid | Delayed Zoledronic Acid
Serious Adverse Events (participants affected / at risk) | 47/254 | 56/269
Other Adverse Events (participants affected / at risk) | 225/254 | 240/269
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Upfront Zoledronic Acid (N=254) | Delayed Zoledronic Acid (N=269)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 3
Angina unstable (Cardiac disorders) | 0 | 1
Bundle branch block left (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 4 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Cytotoxic cardiomyopathy (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 | 0
Goitre (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Cataract cortical (Eye disorders) | 0 | 1
Conjunctival hyperaemia (Eye disorders) | 1 | 0
Corneal oedema (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gingival erosion (Gastrointestinal disorders) | 0 | 1
Gingivitis (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Loose tooth (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 2
Splenic artery aneurysm (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Gait disturbance (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 0
Impaired healing (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Sudden death (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Corneal graft rejection (Immune system disorders) | 1 | 0
Abscess jaw (Infections and infestations) | 1 | 0
Acanthamoeba keratitis (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 1
Breast cellulitis (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 2
Erysipelas (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Pleural infection (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 1
Tooth infection (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 1
Urogenital infection bacterial (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 3
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 2
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Computerised tomogram thorax abnormal (Investigations) | 1 | 0
Weight increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Bone fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 3
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 5
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Primary sequestrum (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amnestic disorder (Nervous system disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Monoplegia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 2
Apathy (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 3
Mental disorder (Psychiatric disorders) | 1 | 1
Mutism (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 3 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 1
Vasoconstriction (Vascular disorders) | 0 | 1
Venous insufficiency (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Upfront Zoledronic Acid (N=254) | Delayed Zoledronic Acid (N=269)
Constipation (Gastrointestinal disorders) | 20 | 16
Nausea (Gastrointestinal disorders) | 24 | 21
Asthenia (General disorders) | 26 | 36
Fatigue (General disorders) | 46 | 57
Influenza like illness (General disorders) | 18 | 5
Oedema peripheral (General disorders) | 20 | 26
Pyrexia (General disorders) | 21 | 3
Bronchitis (Infections and infestations) | 10 | 16
Influenza (Infections and infestations) | 14 | 9
Nasopharyngitis (Infections and infestations) | 12 | 14
Weight increased (Investigations) | 33 | 23
Hypercholesterolaemia (Metabolism and nutrition disorders) | 24 | 33
Arthralgia (Musculoskeletal and connective tissue disorders) | 123 | 136
Back pain (Musculoskeletal and connective tissue disorders) | 41 | 36
Bone pain (Musculoskeletal and connective tissue disorders) | 27 | 21
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 15
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 26 | 34
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 10 | 16
Myalgia (Musculoskeletal and connective tissue disorders) | 33 | 35
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 11 | 18
Pain in extremity (Musculoskeletal and connective tissue disorders) | 26 | 46
Headache (Nervous system disorders) | 24 | 28
Paraesthesia (Nervous system disorders) | 7 | 15
Anxiety (Psychiatric disorders) | 17 | 22
Depression (Psychiatric disorders) | 13 | 24
Insomnia (Psychiatric disorders) | 20 | 11
Vulvovaginal dryness (Reproductive system and breast disorders) | 13 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 17
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 21
Hot flush (Vascular disorders) | 66 | 101
Hypertension (Vascular disorders) | 32 | 25
Lymphoedema (Vascular disorders) | 20 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.